CLINICAL TRIAL: NCT02558166
Title: Relation Between the Renal Resistive Index and Markers of the Systemic Circulation, the Microcirculation, Fluid Status and of Renal Function.
Brief Title: Renal Resistive Index in Patients With Shock
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, H.M. Oudemans-van Straaten, MD, PhD, Prof. Dr., Amsterdam UMC, location VUmc
Other Study IDs: METC-2015.025
Record Dates: First submitted 2015-09-22; First posted 2015-09-23 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Hypovolemic Shock; Cardiogenic Shock; Septic Shock; Kidney Failure, Acute
Keywords: Acute Kidney Injury (AKI); Renal Resistive Index (RRI)
MeSH Terms: conditions — Shock; Shock, Cardiogenic; Shock, Septic; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with shock: Critically ill patients admitted to the intensive care unit (ICU)
  * with shock due sepsis/SIRS, cardiac failure or hemorrhage
  * age > 18 years,
  * noradrenalin support
  * < 24 hours of ICU admission
  * Signed informed consent
- Patients without shock: Critically ill patients admitted to the intensive care unit (ICU)
  * without shock, without vasopressor support and without fluid dependent circulation
  * age > 18 years
  * < 24 hours of ICU admission
  * Signed informed consent

SUMMARY:
This study consists of two substudies.

The first substudy:

'Renal resistive index in critically ill patients with cardiogenic and septic shock'

Design: cross-sectional observational

Aim of this project is:

1. to determine whether critically ill patients with cardiogenic and septic shock have an elevated Renal Resistive Index and
2. to determine whether Renal Resistive Index differs between cardiogenic/hypovolemic shock and shock due to sepsis/systemic inflammation (SIRS)
3. to determine the relation between the (change in) renal vascular resistance and

   * Markers of the systemic - and the microcirculation
   * Fluid status as quantified by bioimpedance analysis
   * Concomitant renal function

The second substudy:

'Predictive value of the Renal Resistive Index on ICU admission and its course for the development of acute kidney injury in critically ill patients with cardiogenic and septic shock'

Design: longitudinal observational

The aim of this project is:

1. to determine whether the renal resistance index on admission to the intensive care unit can predict the development of acute kidney injury (AKI) in critically ill patients with shock
2. to investigate if the renal resistance index on admission to the intensive care unit is an independent predictor of the development of AKI or depends on the severity and duration of shock and other known risk factors of AKI such as comorbidity and use of nephrotoxic drugs

Aim of the large research project is to determine whether the Renal Resistive Index could become a monitoring tool for intervention studies aiming to prevent acute kidney injury or protect the kidney.

DETAILED DESCRIPTION:
Acute Kidney Injury (AKI) is a severe complication developing in intensive care patients as a result of hypovolemic, cardiogenic or septic shock. It is defined by an abrupt decrease in kidney function. It encompasses both direct injury to the kidney as well as acute impairment of function, including decreased glomerular filtration rate (GFR). Its prevention is crucial because AKI increases morbidity and mortality (1). Mechanisms comprise ischemia/reperfusion, oxidative stress, inflammation and toxicity (2).The common pathophysiological pathway includes endothelial damage to microvessels leading to impaired macro- and microvascular flow and this will aggravate ischemia (3).

Up to now, much controversy exists about

* the changes in renal blood flow during different kinds of shock
* the relation between renal blood flow, glomerular filtration rate and the development of AKI
* the relation between renal blood flow and markers of the systemic and microcirculation

In this prospective observational study, three study measurement will be performed in two groups of critically ill patients (shock and no shock).

1. The Renal Resistive Index (RRI) will be determined using Renal Doppler Ultrasound . The renal resistive index (RRI) is a sonographic index assessing resistance of the intrarenal arcuate or interlobar arteries and is used to assess renal arterial disease. It is measured as RRI = (peak systolic velocity - end diastolic velocity)/peak systolic velocity. The normal value is ≈ 0,60, with 0,70 being around the upper limits of normal.
2. The sublingual microcirculation will be quantified using side stream dark field imaging (SDF)
3. Fluid status will be determined by Bioelectrical impedance analysis (BIA) using the Akern device.

In addition, routinely measured markers of circulation, renal function and fluid balance will be collected for analysis.

ELIGIBILITY:
Inclusion Criteria:

First group (patients with shock):

* Critically ill patients admitted to the intensive care unit (ICU) with cardiogenic shock or shock due to sepsis/SIRS or hemorrhage
* Age > 18 years
* Noradrenalin support
* ICU admission < 24 hours
* Signed informed consent

Second group (patients without shock):

* Critically ill patients admitted to the intensive care unit (ICU) without shock, without vasopressor support and without fluid-dependent circulation
* Age > 18 years
* ICU admission < 24-h
* Signed informed consent

In both groups, written consent will be obtained if and when the patients are awake and able to communicate ('deferred consent')

Exclusion Criteria:

* Severe pre-admission chronic renal insufficiency (eGFR < 30 ml/min)
* Dialysis dependency
* Renal transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients, admitted tot the Intensive Care Unit (ICU)
  Variables will be measured in a population of 80 adult patients admitted tot the Intensive Care Unit. This group consists of two groups of 40 patients. The first group consists of 40 patients with cardiogenic or septic shock, the second group will be the control group being intensive care patients without shock. The patients with shock are at increased risk for developing Acute Kidney Injury (AKI).
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2015-08; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
renal resistive index (RRI) | 1 week

SECONDARY OUTCOMES:
Creatine clearance (marker of GFR) | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Heleen M. Oudemans, Prof. Dr., Study Director — Amsterdam UMC, location VUmc
Locations (1):
- VU Medical Center, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Background] Hoste EA, Schurgers M. Epidemiology of acute kidney injury: how big is the problem? Crit Care Med. 2008 Apr;36(4 Suppl):S146-51. doi: 10.1097/CCM.0b013e318168c590. PMID 18382186
- [Background] Basile DP, Anderson MD, Sutton TA. Pathophysiology of acute kidney injury. Compr Physiol. 2012 Apr;2(2):1303-53. doi: 10.1002/cphy.c110041. PMID 23798302
- [Background] Gomez H, Ince C, De Backer D, Pickkers P, Payen D, Hotchkiss J, Kellum JA. A unified theory of sepsis-induced acute kidney injury: inflammation, microcirculatory dysfunction, bioenergetics, and the tubular cell adaptation to injury. Shock. 2014 Jan;41(1):3-11. doi: 10.1097/SHK.0000000000000052. PMID 24346647
- [Background] De Backer D, Orbegozo Cortes D, Donadello K, Vincent JL. Pathophysiology of microcirculatory dysfunction and the pathogenesis of septic shock. Virulence. 2014 Jan 1;5(1):73-9. doi: 10.4161/viru.26482. Epub 2013 Sep 25. PMID 24067428
- [Background] Darmon M, Schortgen F, Vargas F, Liazydi A, Schlemmer B, Brun-Buisson C, Brochard L. Diagnostic accuracy of Doppler renal resistive index for reversibility of acute kidney injury in critically ill patients. Intensive Care Med. 2011 Jan;37(1):68-76. doi: 10.1007/s00134-010-2050-y. Epub 2010 Sep 23. PMID 20862450
- [Background] Schnell D, Deruddre S, Harrois A, Pottecher J, Cosson C, Adoui N, Benhamou D, Vicaut E, Azoulay E, Duranteau J. Renal resistive index better predicts the occurrence of acute kidney injury than cystatin C. Shock. 2012 Dec;38(6):592-7. doi: 10.1097/SHK.0b013e318271a39c. PMID 23042202
- [Background] Dewitte A, Coquin J, Meyssignac B, Joannes-Boyau O, Fleureau C, Roze H, Ripoche J, Janvier G, Combe C, Ouattara A. Doppler resistive index to reflect regulation of renal vascular tone during sepsis and acute kidney injury. Crit Care. 2012 Sep 12;16(5):R165. doi: 10.1186/cc11517. PMID 22971333
- [Derived] Haitsma Mulier JLG, Rozemeijer S, Rottgering JG, Spoelstra-de Man AME, Elbers PWG, Tuinman PR, de Waard MC, Oudemans-van Straaten HM. Renal resistive index as an early predictor and discriminator of acute kidney injury in critically ill patients; A prospective observational cohort study. PLoS One. 2018 Jun 11;13(6):e0197967. doi: 10.1371/journal.pone.0197967. eCollection 2018. PMID 29889830